CLINICAL TRIAL: NCT01929265
Title: A Phase II Study of Bendamustine in Combination With Rituximab as Initial Treatment for Patients With Indolent Non-follicular Non-Hodgkin's Lymphoma
Brief Title: A Phase II Study for Patients With Indolent Non-follicular Non-Hodgkin's Lymphoma
Acronym: IIL INFL09
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIL INFL09
Record Dates: First submitted 2013-08-22; First posted 2013-08-27 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-03

CONDITIONS: Indolent Non-follicular; Non-Hodgkin's Lymphoma
Keywords: INFL; Indolent non-follicular; untreated INFL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Rituximab - Bendamustine (RB) (Experimental): 1 arm: Rituximab - Bendamustine (RB)
  1 arm for all patients
  Interventions: Drug: Bendamustine

INTERVENTIONS:
Drug: Bendamustine — INDUCTION PHASE
  Rituximab - Bendamustine (RB): cycles 1 to 4 (0, 4, 8, 12 week):
  Rituximab: 375 mg/sqm iv, day 1*
  Bendamustine: 90 mg/sqm iv, days 1-2 or days 2-3 according to istitutional/patient/physician choice
  Repeat cycles every 28 days for a total of 4 cycles
  *In cycle 1, in order to avoid tumor lysis syndrome, Rituximab will be given on day 8.
  CONSOLIDATION PHASE
  Rituximab - Bendamustine (RB): cycles 5 to 6 (16, 20 week):
  Rituximab: 375 mg/sqm iv day 1
  Bendamustine: 90 mg/sqm iv days 1-2 or days 2-3 according to istitutional/patient/physician choice
  Rituximab two monthly doses
  Rituximab: 375 mg/sqm iv week 24 and 28
  Other Names: RIBOMUSTIN

SUMMARY:
This is a prospective, multicenter phase II trial designed to determine efficacy and safety of a chemoimmunotherapy with the combination of Bendamustine + Rituximab in patients with advanced untreated Indolent non Follicular non-Hodgkin Lymphomas (INFL).

DETAILED DESCRIPTION:
This is a prospective, multicenter phase II trial designed to determine efficacy and safety of a chemoimmunotherapy with the combination of Bendamustine + Rituximab in patients with advanced untreated Indolent non Follicular non-Hodgkin Lymphomas (INFL).

The study includes and induction phase and a consolidation phase.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent form
2. Histological (bone marrow or lymph nodes biopsy) proven diagnosis of B-cell CD20- positive non-follicular NHL according to REAL/WHO Classification:

   i. small lymphocytic lymphoma-SLL (bone marrow or lymph nodes biopsy ii. lymphoplasmacytic/citoid lymphoma/ Waldenstrom macroglobulinemia(bone marrow or lymph nodes biopsy) iii. nodal marginal zone lymphoma (lymph nodes biopsy)
3. Untreated patients
4. Stage III or IV or stage II with more than three involved sites
5. Presence of at least one of the following criteria for the definition of active disease:

   1. Systemic symptoms
   2. Hemoglobin less than 10 g/dL (due to lymphoma)
   3. Platelets less than 100 x 10 9/L (due to lymphoma)
   4. Diffuse bone marrow infiltrate
   5. Lymphocyte doubling time less than 12 months (in leukemic cases)
   6. Bulky disease (>7 cm)
6. Aged 18 - 75 Life expectancy >6 months
7. ECOG performance status 0-2
8. LVEF ≥45% or FS ≥37%
9. ANC ≥1 x 10 9/l and Platelets count ≥75 x 10 9/l, unless due to bone marrow involvement by follicular lymphoma
10. Creatinine up to 1.5 x ULN
11. Conjugated bilirubin up to 2 x ULN
12. Alkaline phosphatase and transaminases up to 2 x ULN
13. Written informed content

Exclusion Criteria:

1. Patients with diagnosis of marginal zone lymphoma of splenic or MALT origin
2. Patients with diagnosis of typical Chronic Lymphocytic Leukemia (CLL)
3. Men not agreeing to take adequate contraceptive precautions during and for at least 6 months after cessation of therapy
4. History of other malignancies within 3 years prior to study entry except for: adequately treated carcinoma in situ of the cervix; basal or squamous cell skin cancer; low grade, early stage, localized prostate cancer treated surgically with curative intent; good prognosis DCIS of the breast treated with lumpectomy alone with curative intent
5. Medical condition requiring long term use (>1 months) of systemic corticosteroids
6. Active bacterial, viral, or fungal infection requiring systemic therapy
7. Concurrent medical condition which might exclude administration of therapy
8. Cardiac insufficiency (NYHA grade III/IV)
9. Myocardial infarction within 6 months of entry on study
10. Severe chronic obstructive pulmonary disease with hypoxemia
11. Severe diabetes mellitus difficult to control with adequate insulin therapy
12. Hypertension that is difficult to control
13. Impaired renal function with creatinine clearance <30 ml/min
14. HIV positivity
15. HBV positivity with the exception of patients HbsAg negative and Ab anti-Hbcore positive(these patientes need to receive prophylaxis with Lamivudine)
16. HCV positivity with the exception of patients with HCV RNA negative.
17. CNS involvement by lymphoma
18. Participation at the same time in another study in with investiogational drugs are used
19. Known hypersensitivity or anaphylactic reactions to murine antibodies or proteins
20. Any other co-existing medical or psychological condition that would preclude participation in the study or compromise ability to give informed consent
21. Women in pregnancy or breastfeeding

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2011-01; Primary Completion 2012-03 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Complete remission rate (CR) | 5 months
  Evaluated at the end of treatment

SECONDARY OUTCOMES:
Safety analysis | 5 months
  Evaluated during and at the end of treatment. Percentage of patients with adverse, hematological and non-hematological toxic events
Overall response rate (ORR) | 5 months
  Evaluated at the end of treatment. Complete plus partial remission.
Overall survival (OS) | at 2 years
  Dead for any causes after diagnosis. Evaluated by means of Kaplan-Meier method.
Progression free survival (PFS) | at 2 years
  Progression, relapse or dead for any causes after diagnosis. Evaluated by means of Kaplan-Meier method.
Disease free survival (PFS) | at 2 years
  Relapse or dead for any causes from the end of treatment, for patients in CR after B+R. Evaluated by means of Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Luca Baldini, Prof., Principal Investigator — UOC Ematologia 1/CTMO, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico
Locations (25):
- Italy (25):
  - SC Ematologia - AO SS. Antonio e Biagio e C. Arrigo, Alessandria, AL
  - SC Ematologia Spedali Civili, Brescia, BS
  - Divisione di Ematologia e Trapianti, Ospedale San Maurizio, Bolzano, BZ
  - Divisione di Ematologia, Centro Trapianto di Cellule Staminali, San Giovanni Rotondo, Foggia
  - Divisione Ematologia I , Ospedale San Martino, Genova, GE
  - S.C. Ematologia Azienda Ospedaliera Papardo, Messina, ME
  - Divisione di Oncologia Medica ed Ematologia, Istituto Clinico Humanitas, Rozzano, Milano
  - Divisione di Ematologia Ospedale Niguarda, Milan, MI
  - Centro Oncologico Modenese, Modena, MO
  - Ematologia Azienda Ospedaliero Universitaria Paolo Giaccone, Palermo, PA
  - Div. Oncologia Medica - CRO, Centro di Riferimento Oncologico, Aviano, PN
  - UOC Ematologia 1/CTMO, Fondazione IRCCS Cà Granda Ospedale Maggiore Policlinico, Milan
  - Oncoematologia Istituto Pascale, Napoli
  - S.C.D.U Ematologia Azienda Ospedaliero Universitaria Maggiore, Novara
  - UO Ematologia Università - Policlinico San Matteo, Pavia
  - Ematologia Ospedale Santo Spirito, Pescara
  - UOA Ematologia, Ospedale Civile Ospedale G. da Saliceto, Piacenza
  - Div. Ematologia AO Bianchi Melacrino Morelli, Reggio Calabria
  - Ematologia, Azienda Ospedaliera Arcispedale "S.Maria Nuova", Reggio Emilia
  - Ematologia, Università "La Sapienza", Roma
  - Clinica Ematologia Policlino Le Scotte, Siena
  - Struttura Complessa di Onco-Ematologia Azienda Ospedaliera S.Maria, Terni
  - SC Ematologia - Città della Salute e della Scienza, Torino
  - SC Ematologia U - Città della Salute e della Scienza, Torino
  - Clinica Ematologica e Unità di Terapie Cellulari 'Carlo Melzi' AOU S. Maria della Misericordia, Udine